CLINICAL TRIAL: NCT01883349
Title: Cognitive Impairment and Imaging Correlates in End Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13566
Record Dates: First submitted 2013-05-30; First posted 2013-06-21 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ESRD patients: ESRD patients awaiting renal transplantation
  Interventions: Procedure: Kidney Transplant
- Control Arm: Subjects without kidney disease. No intervention with control group.
  Interventions: Other: No kidney transplant

INTERVENTIONS:
Procedure: Kidney Transplant — Kidney Transplant Surgery
  Groups: ESRD patients
Other: No kidney transplant — The control group was made up of subjects without ESRD and were not on the renal transplantation waitlist.
  Groups: Control Arm

SUMMARY:
This is an observational cohort to understand cognitive impairment in end stage renal disease before and after a kidney transplant.

DETAILED DESCRIPTION:
Cognitive impairment is very common in patients with End Stage Renal Disease (ESRD). It exact mechanisms are not clear, but patients with ESRD have more cerebral white matter changes. Several studies have shown that cognitive function improves post-transplant, indicating that there may be some reversibility in the process. This study will examine the correlation between cognitive impairment and structural brain changes before and after renal transplantation. We will also study the correlation of cognitive function with serum inflammatory markers before and after transplant. These results will be compared to aged matched healthy controls without kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Pre-transplant ESRD patients who are listed for renal transplantation
* Able to sign pre-transplant consent on their own will
* Have english as their native language

Exclusion Criteria:

* Current use of antipsychotics or anti-epileptics
* Inability to read or write which will limit their ability to perform the cognitive tests
* Claustrophobia or inability to get MRI for other reasons
* Unable to sign consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients from the renal transplant waiting list at University of Kansas Medical Center. They will be tested before renal transplant and 3 months and 12 months after renal transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2023-07 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  Cognition will be assessed using relevant neuropsychological tests used by National Alzheimers Coordination center (NACC) uniform data set (UDS). Primary outcome will be logical memory. Score range 0-25. Higher scores indicate better cognitive function.

SECONDARY OUTCOMES:
Change in brain MRI | Change from Baseline to 3 Months and 12 months after Renal Transplant
  Brain MRI will be performed before and after transplant
Change in inflammatory markers | Change from Baseline to 3 months and 12 months post transplant
Change in verbal declarative/episodic memory | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  WMS-R Logical Memory I- Immediate is a test where a brief story is read to subject, who is then asked to retell it from memory immediately; primary measure of performance is number of story units recalled. Scores are from 0-25 with higher scores indicating better cognition.
Change in delayed verbal declarative/episodic memory | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  WMS-R Logical Memory II- Delayed measures delayed recall of story read to the participant at the beginning of testing session (WMS-R Logical Memory I- Immediate). Scores range from 0-25 with higher scores indicating better cognition.
Change in psychomotor speed and visuospatial function | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  WAIS-R Digit Symbol Substitution test is where a subject is given a key consisting of numbers 1-9, each paired with a unique, easy-to-draw symbol; subject fills in corresponding symbol for each number in a limited time. Scores are from 0-133 with higher scores indicating better cognition.
Change in general dementia screening score | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  Mini-Mental State Examination Screening scale evaluates orientation to place, orientation to time, registration, attention and concentration, recall, language, and visual construction. Scores range from 0-30 with higher scores indicate better cognition.
Change in working memory or attention | Change from Baseline to 3 Months and 12 Months after Renal Transplant
  Digit Span forward and backward are tests where a subject is read sequences of increasing length and asked to repeat them. Digit span length is the length of the highest digit sequence the subject is able to repeat correctly. Scores range from 0-12 with higher scores indicate better cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Gupta, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Lepping RJ, Montgomery RN, Sharma P, Mahnken JD, Vidoni ED, Choi IY, Sarnak MJ, Brooks WM, Burns JM, Gupta A. Normalization of Cerebral Blood Flow, Neurochemicals, and White Matter Integrity after Kidney Transplantation. J Am Soc Nephrol. 2021 Jan;32(1):177-187. doi: 10.1681/ASN.2020050584. Epub 2020 Oct 16. PMID 33067382
- [Result] Gupta A, Lepping RJ, Yu AS, Perea RD, Honea RA, Johnson DK, Brooks WM, Burns JM. Cognitive Function and White Matter Changes Associated with Renal Transplantation. Am J Nephrol. 2016;43(1):50-7. doi: 10.1159/000444334. Epub 2016 Feb 20. PMID 26894920